CLINICAL TRIAL: NCT07314398
Title: Prospective Cohort Study on Surgical Methods and Outcomes in Emergency Groin and Ventral Hernia Repairs in Finland
Brief Title: Emergency Hernia Repair
Status: Not yet recruiting | Type: Observational
Sponsor: Oulu University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 50/2023
Record Dates: First submitted 2025-09-01; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-10

CONDITIONS: Emergency Inguinal Hernia Repair; Emergency Ventral Hernia Repair
Keywords: inguinal hernia; ventral hernia; emergency surgery
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency ventral or inguinal hernia repair: Patients, who will have their ventral or inguinal hernia repaired in emergency surgery
  Interventions: Procedure: Emergency hernia repair

INTERVENTIONS:
Procedure: Emergency hernia repair — Patients who will have either their ventral or inguinal hernia repaired in emergency surgery. The techniques are not standardized, but the details will be collected to prospective database.

SUMMARY:
Emergency hernia repairs are associated with significantly higher morbidity and mortality compared with elective hernia surgery. In Finland, approximately 500 emergency groin hernia repairs and 600 ventral hernia repairs are performed annually, but treatment practices vary widely, and high-quality evidence is lacking.

This prospective multicenter cohort study will evaluate outcomes of emergency groin and ventral hernia repairs in Finland. About 600 patients will be recruited over two years and followed for five years postoperatively. The study will collect standardized data on patient demographics, comorbidities, surgical technique, intraoperative findings, postoperative course, and long-term follow-up. Quality of life will be assessed with RAND-36, AAS, and PROMIS questionnaires.

The primary endpoint is hernia recurrence within two years after surgery. Secondary outcomes include 30- and 90-day complications, infection rates, readmissions, recovery time, and quality of life at 1, 2, and 5 years.

The results will provide robust evidence to guide clinical practice, optimize surgical techniques, and refine urgency classification and surgeon competence requirements for emergency hernia repair.

DETAILED DESCRIPTION:
1. Introduction and Background

   Hernia surgery is among the most common surgical procedures, the majority performed as elective operations. However, the proportion of emergency procedures is considerable, and these are associated with significantly higher morbidity and mortality compared with elective surgery.

   In Finland, approximately 500 emergency groin hernia repairs and 600 ventral hernia repairs are performed annually. Current treatment practices for emergency hernia surgery vary substantially, and scientific evidence on management and outcomes is lacking. Existing guidelines are partly outdated and largely based on expert opinion.

   The aim of this study is to provide new, scientifically robust evidence on the outcomes, complications, and postoperative quality of life following emergency hernia surgery.
2. Study Objectives

   The primary objective is to assess the short- and long-term outcomes of different surgical techniques in emergency groin and ventral hernia repairs. Specifically, the study will evaluate:

   Surgical outcomes and complications within 30 and 90 days postoperatively

   Risk of recurrence and quality of life at 1, 2, and 5 years

   Impact of wound and mesh infections, as well as other postoperative factors, on recurrence

   Effectiveness and safety of different surgical techniques

   The results will support more evidence-based and precise recommendations on surgical methods, urgency classification, and the role of surgeon expertise.
3. Study Design and Patient Cohort

   This is a multicenter study with a prospective patient cohort of emergency groin and ventral hernia repairs. Patients will be recruited over two years and followed up for five years postoperatively. The aim is to include as many eligible patients as possible.

   Inclusion criterion

   Emergency repair of a groin or ventral hernia

   Exclusion criteria

   Pregnancy

   Age under 18 years

   Advanced malignancy

   Inability to follow up (e.g., long travel distance or poor functional status)

   Participation in another study

   Lack of informed consent

   Estimated sample size: ~600 patients recruited across participating Finnish hospitals.
4. Methods and Data Collection

   Data will be collected in the REDCap system at the following time points:

   Baseline (preoperative): Patient demographics (age, sex, BMI) and comorbidities

   Intraoperative: Surgical technique, procedures performed, duration of surgery

   Postoperative (hospital stay): Recovery, complications, reoperations

   Follow-up at 30 days, 90 days, 1, 2, and 5 years:

   Recurrence (clinically and with imaging if needed)

   Quality of life (RAND-36, AAS, PROMIS)

   Complications, readmissions, recovery time, sick leave

   Patients will be contacted by phone at each follow-up. If recovery is delayed, complications are suspected, or recurrence is possible, patients will be invited for further assessment at the hospital where the surgery was performed.
5. Statistical Analysis

   The primary endpoint is hernia recurrence within two years after surgery.

   Statistical methods include:

   Kaplan-Meier analysis for comparison of surgical techniques

   Chi-square test and Fisher's exact test for categorical variables

   Student's t-test for continuous variables

   Multivariate analysis for independent risk factors

   Analyses will be conducted using IBM SPSS Statistics. A p-value < 0.05 will be considered statistically significant.
6. Ethical Considerations and Data Protection

   The study has been approved by the Ethics Committee of the Wellbeing Services County of North Ostrobothnia. Local research permits will be obtained from each participating hospital before study initiation.

   Participation is voluntary, and written informed consent will be obtained from all patients. Clinical management will follow local treatment protocols regardless of study participation. Patient data will be stored in a pseudonymized form. The data controller is the Wellbeing Services County of North Ostrobothnia.
7. Timeline

2024-2026: Patient recruitment and initiation of follow-up. Study start date: 1 September 2025 across all participating hospitals.

2028: Data analysis and first publication on the primary endpoint

2031: Completion of follow-up and publication of long-term outcomes

ELIGIBILITY:
Inclusion Criteria:

* Emergency repair of a groin or ventral hernia

Exclusion Criteria:

* Pregnancy
* Age under 18 years
* Advanced malignancy
* Inability to follow up (e.g., long travel distance or poor functional status)
* Participation in another study
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, who will undergo emergency ventral or inguinal hernia repair between Oct 1st 2025 and Sep 31st 2027 in participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with hernia recurrence | 2 years
  Either clinical or radiological recurrent hernia
  * Risk of recurrence and quality of life at 1, 2, and 5 years
  * Impact of wound and mesh infections, as well as other postoperative factors, on recurrence
  * Effectiveness and safety of different surgical techniques

SECONDARY OUTCOMES:
Surgical site infection rate 30 days after surgery | 30 days
  Surgical site infection as described by Centers for Disease Control and Prevention
Incidence of Postoperative complications 30 after the surgery | 30 days
  Surgical complications graded by Clavien-Dindo Classification
Number of patients who died 30 days after the surgery | 30 days
  Death after the surgery
Incidence of hernia related re-operations during the 5 years' follow-up | 5 years
  Reoperations due to recurrent hernia, mesh or other operations at the previous hernia site
Quality of life RAND-36 | 5 years
  Quality of life measured by RAND-36
Quality of life Activities Assessment Scale | 5 years
  Quality of life measured by Activities Assessment Scale
Quality of life PROMIS | 5 years
  Quality of life measured by promis

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due to Finnish laws on privacy protection but are available from the corresponding author on reasonable request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT07314398/Prot_SAP_000.pdf